CLINICAL TRIAL: NCT02123108
Title: Safety and Efficacy of Basiliximab, Delayed Dose Tacrolimus Plus ECMPA, Versus Standard Dose Tacrolimus, ECMPA Plus Corticosteroids in Patients Undergoing Liver Transplant
Brief Title: Safety and Efficacy of Basiliximab, Delayed Dose Tacrolimus Plus ECMPA (Enteric Coated Mycophenolic Acid) Following Liver Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Fady M Kaldas, M.D., F.A.C.S., Principle-Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCLA: CCHI621AUS17T
Record Dates: First submitted 2014-02-24; First posted 2014-04-25 (Estimated); Results first posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Liver Transplantation
Keywords: Simulect; Myfortic; Orthotopic liver transplantation (OLT); Renal Dysfunction
MeSH Terms: conditions — Renal Insufficiency | interventions — Basiliximab; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basiliximab (Experimental): Tacrolimus with Basiliximab induction
  Interventions: Drug: Basiliximab; Drug: Tacrolimus; Drug: Mycophenolic Acid
- Tacrolimus Group (Active Comparator): Tacrolimus (without basiliximab induction); standard of care group
  Interventions: Drug: Tacrolimus; Drug: Mycophenolic Acid

INTERVENTIONS:
Drug: Basiliximab — Peri-operative 40 mg IV dose within 4 hours of OLT Postoperative 20mg IV dose Day 4
  Other Names: Simulect
  Arms: Basiliximab
Drug: Tacrolimus — Day #7 post-transplant or when serum creatinine (SCr) < 1.8 mg/dl 6 months to 1 year: 0.03-0.1 mg.kg q12h po to maintain whole blood trough concentration of 3-5ng/mL
  Other Names: Prograf
  Arms: Basiliximab
Drug: Tacrolimus — Day #1 post-transplant to 6 months: 0.03-0.1mg/kg q12h po to maintain whole blood trough concentration of 7-10 ng/mL + 6 months to 1 year: maintain whole blood trough concentration of 5-8ng/mL
  Other Names: Prograf
  Arms: Tacrolimus Group
Drug: Mycophenolic Acid — Enteric coated mycophenolic acid 360-720 mg po bid
  Other Names: Myfortic; Mycophenolate sodium

SUMMARY:
This is an investigator initiated study at the University of California, Los Angeles (UCLA) funded by Novartis looking at using a combination of immunosuppressive drugs in liver transplant patients that are at risk of developing kidney problems. Kidney problems following liver transplants is the most problematic issue facing liver transplant patients today.

This study will generate information in this area of high unmet medical need utilizing basiliximab and Myfortic and using a reduced dose of tacrolimus, one of the current standard of care medications, after kidney function has normalized.

DETAILED DESCRIPTION:
Since basiliximab works on the same receptor system as tacrolimus and has not been shown to cause significant adverse effects, such as nephrotoxicity or the cytokine release syndrome, the investigators are proposing induction therapy with basiliximab in liver transplant patients with concomitant preoperative renal dysfunction. This will combat acute rejection and allow the delay of tacrolimus therapy until post-operative day #7. The delay in tacrolimus therapy should allow renal function to improve and reduce the chance of continued renal dysfunction. Also, the addition of basiliximab to the immunosuppressive regimen should allow for a reduction in tacrolimus dose (normal tacrolimus concentrations at UCLA are 7-10ng/mL. Our goal will be 3-5ng/mL) in the immediate post-transplant period thereby reducing the chance of acute and long-term efficacy-limiting adverse effects associated with the tacrolimus while maintaining adequate immunosuppression to reduce acute rejection episodes. This would be the most convincing prospective randomized study utilizing basiliximab as a renal sparing agent in liver transplantation.

Objectives Primary objectives

• To evaluate renal recovery/ function following OLT in patients undergoing orthotopic liver transplant at 6 and 12 months post-transplant.

Secondary objectives (comparing the two treatment arms)

* To determine the tolerability and adverse event profile during the first year post-transplant.
* To determine incidence and severity acute rejection episodes
* To determine the incidence of death and/or graft failure within the first year post-transplant

Study design The study is a single center prospective randomized trial wherein the investigators will have two groups. Patients will be screened and eligible patients will be enrolled pre-transplant. Patients will then be randomized at time of transplant to either the control or treatment arm. Post transplant laboratory data (chemistry, tacrolimus level and liver function tests) will be collected on a daily basis. For the duration of the patients' hospital stay (average 2-3 weeks). This will provide the early data set for early post operative results. Patients will subsequently be followed on a weekly outpatient basis upon discharge as per protocol. During these visits, laboratory data (chemistry, tacrolimus level and liver function tests) are also collected and will provide the continued flow of data for our follow up analysis. Any evidence of rejection will prompt treatment with rescue therapy and if necessary disenrollment from the study.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfill all of the following criteria:

* >18 years old
* Undergoing first or second OLT
* MELD (model for end-stage liver disease) score >25
* Serum creatinine > 1.5 or ongoing hemodialysis for less than 4 weeks at the time of transplant
* Able and agreeable to conform to requirements of the study
* Patients or proxy must give written informed consent before any assessment is performed.

Exclusion Criteria:

* <18 years old
* Serum creatinine <1.5
* MELD Score < 25
* Ongoing hemodialysis for 4 or more weeks (those patients become eligible for renal transplants at that point per UCLA practice).
* Receiving OKT3 (Muromonab-CD3), ATG (Antithymocyte Globulin), or IVIG (Intravenous Immunoglobulin Therapy) therapy around time of transplant
* Participating in another clinical research study involving the evaluation of another investigational drug or device
* Prior documented allergy to any of the study medications
* Active Fungal infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fady M Kaldas, MD, Principal Investigator — UCLA Department of Surgery
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramirez CB, Marino IR. The role of basiliximab induction therapy in organ transplantation. Expert Opin Biol Ther. 2007 Jan;7(1):137-48. doi: 10.1517/14712598.7.1.137. PMID 17150025
- [Background] Katari SR, Magnone M, Shapiro R, Jordan M, Scantlebury V, Vivas C, Gritsch A, McCauley J, Starzl T, Demetris AJ, Randhawa PS. Clinical features of acute reversible tacrolimus (FK 506) nephrotoxicity in kidney transplant recipients. Clin Transplant. 1997 Jun;11(3):237-42. PMID 9193849
- [Background] Rimola A, Gavaler JS, Schade RR, el-Lankany S, Starzl TE, Van Thiel DH. Effects of renal impairment on liver transplantation. Gastroenterology. 1987 Jul;93(1):148-56. doi: 10.1016/0016-5085(87)90327-1. PMID 3556303
- [Background] Klintmalm GB, Gonwa TA. Nephrotoxicity associated with cyclosporine and FK506. Liver Transpl Surg. 1995 Sep;1(5 Suppl 1):11-9. PMID 9346596
- [Background] Guckelberger O, Bechstein WO, Neuhaus R, Luesebrink R, Lemmens HP, Kratschmer B, Jonas S, Neuhaus PL. Cardiovascular risk factors in long-term follow-up after orthotopic liver transplantation. Clin Transplant. 1997 Feb;11(1):60-5. PMID 9067697
- [Background] Neuhaus P, Clavien PA, Kittur D, Salizzoni M, Rimola A, Abeywickrama K, Ortmann E, Chodoff L, Hall M, Korn A, Nashan B; CHIC 304 International Liver Study Group. Improved treatment response with basiliximab immunoprophylaxis after liver transplantation: results from a double-blind randomized placebo-controlled trial. Liver Transpl. 2002 Feb;8(2):132-42. doi: 10.1053/jlts.2002.30302. PMID 11862589
- [Background] Calmus Y, Scheele JR, Gonzalez-Pinto I, Jaurrieta EJ, Klar E, Pageaux GP, Scudamore CH, Cuervas-Mons V, Metselaar HJ, Prestele H, Girault D. Immunoprophylaxis with basiliximab, a chimeric anti-interleukin-2 receptor monoclonal antibody, in combination with azathioprine-containing triple therapy in liver transplant recipients. Liver Transpl. 2002 Feb;8(2):123-31. doi: 10.1053/jlts.2002.30882. PMID 11862588
- [Background] Onrust SV, Wiseman LR. Basiliximab. Drugs. 1999 Feb;57(2):207-13; discussion 214. doi: 10.2165/00003495-199957020-00006. PMID 10188761
- [Background] Cherqui D, Duvoux C, Charlotte F, Humeres R, Lauzet JY, Metreau JM, Salvat A, Rotman N, Julien M, Fagniez PL, et al. [Value of a powerful initial immunosuppression after liver transplantation. Prospective study of 60 cases]. Gastroenterol Clin Biol. 1994;18(2):115-22. French. PMID 8013792
- [Background] Berard JL, Velez RL, Freeman RB, Tsunoda SM. A review of interleukin-2 receptor antagonists in solid organ transplantation. Pharmacotherapy. 1999 Oct;19(10):1127-37. doi: 10.1592/phco.19.15.1127.30582. PMID 10512062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Basiliximab | Tacrolimus Group
Started | 30 | 29
Completed | 28 | 26
Not Completed | 2 | 3
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basiliximab | Tacrolimus Group | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Full Range); unit: years] | 59 [25 to 70] | 56.7 [25 to 70] | 57.9 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 21 | 32
  Male | 19 | 8 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Renal Recovery/ Function
Description: Number of participants who experienced dialysis independence or improvement based upon kidney function labs as a measure of renal recovery/ function following OLT in patients after undergoing orthotopic liver transplant
Time Frame: 12 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Basiliximab | Tacrolimus Group
Number analyzed (Participants) | 28 | 26
Participants | 28 | 26

2. Other Pre Specified Outcome: Participants Experiencing Adverse Event Attributable to Study Drug
Time Frame: 12 months post liver transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Basiliximab | Tacrolimus Group
Number analyzed (Participants) | 30 | 29
Participants | 0 | 0

3. Other Pre Specified Outcome: Participants Experiencing Acute Rejection Episode
Time Frame: 12 months post liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Basiliximab | Tacrolimus Group
Number analyzed (Participants) | 30 | 29
Participants | 3 | 4

4. Other Pre Specified Outcome: Survival
Description: Participants at risk minus incidence of death within the first year post-transplant
Time Frame: 12 months post liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Basiliximab | Tacrolimus Group
Number analyzed (Participants) | 30 | 29
Participants | 28 | 26

5. Other Pre Specified Outcome: Participants Experiencing Graft Failure
Time Frame: 12 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Basiliximab | Tacrolimus Group
Number analyzed (Participants) | 30 | 29
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Basiliximab | Tacrolimus Group
All-Cause Mortality (participants affected / at risk) | 2/30 | 3/29
Serious Adverse Events (participants affected / at risk) | 2/30 | 3/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basiliximab (N=30) | Tacrolimus Group (N=29)
Death (General disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes